CLINICAL TRIAL: NCT06769256
Title: Effects of Intracoronary Recombinant Human TNK Tissue-type Plasminogen Activator Versus Tirofiban on Myocardial Perfusion and Clinical Prognosis in Patients With ST-segment Elevation Myocardial Infarction and High Thrombus Burden: a Multicenter, Randomized, Controlled, Single-blind, Non-inferior Study
Brief Title: Intracoronary rhTNK-tPA Versus Tirofiban in Patients With STEMI and High Thrombus Burden
Acronym: H2-THROMBUS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Principal Investigator, Chuanyu Gao, Director, Henan Institute of Cardiovascular Epidemiology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HenanICE202412
Record Dates: First submitted 2024-12-26; First posted 2025-01-10 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Tirofiban

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracoronary rhTNK-tPA (Experimental)
  Interventions: Drug: rhTNK-tPA, 4-8 mg
- Intracoronary Tirofiban (Active Comparator)
  Interventions: Drug: Tirofiban

INTERVENTIONS:
Drug: rhTNK-tPA, 4-8 mg — Intracoronary influsion of rhTNK-tPA (4 mg). After 10 minutes of administration, 4 mg may be given again if the thrombus burden is not significantly reduced.
  Arms: Intracoronary rhTNK-tPA
Drug: Tirofiban — Intracoronary influsion of Tirofiban (10 µg/kg) , and then administered intravenously at 0.075-0.15 µg/kg.min for 36 h or longer
  Arms: Intracoronary Tirofiban

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of intracoronary rhTNK-tPA or Tirofiban in patients with ST-segment elevation myocardial infarction and high thrombus burden. The main questions it aims to answer are:

* Is the efficacy of intracoronary rhTNK-tPA non-inferior to intracoronary Tirofiban for the treatment of ST-segment elevation myocardial infarction in patients wiht high thrombus burden?
* Does intracoronary rhTNK-tPA increase the incidence of bleeding events?

This multicenter RCT study plans to enroll 300 patients, who are randomly divided into two groups: intracoronary rhTNK-tPA or Tirofiban by 1:1. The primary efficacy endpoint was post-PCI corrected TIMI frame count (CTFC). Major adverse events (death, recurrent myocardial infarction, ischemic stroke, or hospitalization for heart failure) were observed at 1 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old;
* STEMI within 12 hours of onset;
* TIMI flow grade 0-2 or TIMI thrombus grade ≥4 after thrombus aspiration or balloon dilation
* Radial artery access

Exclusion Criteria:

* A functional coronary collateral supply (Rentrop grade≥2) to the infarctrelated artery
* Known or suspected old myocardial infarction of target vessels
* Rescue PCI
* Cardiogenic shock
* Contraindications to Tirofiban or rhTNK-tPA
* Severe hepatic and renal insufficiency (alanine aminotransferase ≥5 upper limit of normal; estimated glomerular filtration rate <30ml/min/1.73m2, or on dialysis)
* Prolonged (> 10 minutes) cardiopulmonary resuscitation
* Definite mechanical complications (including ventricular septal perforation, or rupture of the Papillary tendon bundle, or rupture of the left ventricular free wall)
* Severe chronic obstructive pulmonary disease or respiratory failure
* Severe infection
* Neurological disorders
* Malignant tumors or other pathophysiological conditions with an expected survival time of less than 1 year
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Corrected TIMI frame count (CTFC) | At the end of Percutaneous Coronary Intervention procedure

SECONDARY OUTCOMES:
TIMI flow grade | At the end of Percutaneous Coronary Intervention procedure
Complete ST-segment resolution (STR) | 1 hour post PCI procedure
Left ventricular ejection fraction (LVEF) | Baseline, 1 month, 6 months and 12 months
A composite of all-cause death, recurrent myocardial infarction, ischemic stroke, and hospitalization for heart failure | 1 month, 6 months and 12 months
Bleeding events according to the BARC bleeding classification | At hospital discharge, an average of 2 days after primary PCI, 1 month, 6 months and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan, China